CLINICAL TRIAL: NCT03351959
Title: Complete Pathologic Response Rectal Cancers EYSAC.1 Study
Brief Title: Complete Pathologic Response Rectal Cancers
Acronym: CORSiCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: European Society of Surgical Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: FPAG002
Record Dates: First submitted 2017-11-14; First posted 2017-11-24 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2017-11

CONDITIONS: Rectal Cancer
Keywords: ypT0
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ypT0 rectal cancers: Rectal cancer patients who underwent neo-adjuvant treatment followed by surgical resection and had a final pathologic diagnosis of absence of residual viable tumoral cells within the rectal wall specimen (pathologic complete response, pCR - ypT0).
  Interventions: Radiation: neo-adjuvant treatment

INTERVENTIONS:
Radiation: neo-adjuvant treatment — long-course radio-chemoradiation; short-course radiation with immediate/delayed surgery

SUMMARY:
Background. About 20% of rectal cancers who underwent neoadjuvant treatment (neoCHT-RT) achieve a pathological complete response in the surgical specimen(ypT0); however, about 10% of ypT0 present metastatic nodes (N+). Although seldom analyzed, ypT0N+ identification could be crucial in order to tailor treatments.

Hypotheses. The two hypotheses to test are if we can identify ypT0N+ and if N+ is an independent prognostic factor.

Aim 1. To create a large Database (DB) of ypT0. Aim 2. To compare ypT0N0 vs ypT0N+ with respect of their clinical/radiological/molecular features.

Aim 3. To investigate long term results. Preliminary Study. Dr Lorenzon is the PI of an Italian retrospective multicentric study conducted on 260 ypT0 focused on treatment and outcomes.

Design. The PI will operate in partnership with the European Society of Surgical Oncology (ESSO). A DB will be used by ESSO-affiliated centres for collecting the clinical, pathological and radiological data of ypT0N0/N+, previously treated (last 5 years) and prospectively enrolled (6 months + 2 years of follow-up); each centre will provide a junior (<40 yrs) member for data collection and a senior investigator .for data validation; all the analyses will be centralized by the PI. ypT0N0 and ypT0N+ will be compared for the clinical/pathological variables, for the gene expression profiles of pre-neoCHT-RT biopsies (grant requested). Uni-multivariate survival analyses (end-points: OS, DFS, DSS) will be conducted at 2 years of follow-up.

Impact. This is the first study aimed to investigate ypT0N+ features; their accurate identification could lead to treat safely thousands of ypT0N0/year with local excisions leaving major surgery for N+ patients. Results will change practice and reduce considerably health-related costs; moreover, the molecular profiles will open new frontiers of research.

DETAILED DESCRIPTION:
Prospectus. The COmplete pathologic ReSponse rectal Cancers EYSAC.1 Study (CORSiCA) proposed by Dr Lorenzon will be conducted at the Fondazione Policlinico Universitario Agostino Gemelli in Rome in partnership with the European Society of Surgical Oncology (ESSO) - Young Alumni Club, and it will focus on rectal cancer patients who underwent neo-adjuvant treatment followed by surgical resection and had a final pathologic diagnosis of absence of residual viable tumoral cells within the rectal wall specimen (pathologic complete response, pCR - ypT0).

Background. With about 135.000 new European cases each year, rectal cancer is a major European issue representing also a field of major investigations. Indeed, over the last 3 decades important advances have been made in the clinical/surgical management of these patients: the most significant ones were the introduction of total mesorectal excision (TME) and the use of neo-adjuvant (chemo)radiation treatments (neoCHT-RT) which changed dramatically the state of art and the multimodal approach to this disease. Currently, the latest international guidelines recommend performing a neoCHT-RT in locally advanced, non-metastatic rectal cancers, clinically staged as ≥T3 any N, anyT N+ or if the circumferential resection margin (CRM) is less than 1 mm, since this approach results in less local recurrences, tumor down-sizing and down-staging. In line with all the improvements made so far, the ultimate effect of neoCHT-RT is the achievement of a complete response, which may be defined as clinical (absence of residual primary tumor clinically detectable, cT0) or pathological. ypT0 occurs in about 20% of patients who underwent neoCHT-RT. Of note, neoadjuvant treatment modalities include a short-course radiotherapy (short RT) followed by immediate surgery or a long course chemo-radiotherapy (CHT-RT) followed by surgery delayed after an interval of at least 4 weeks. Literature about complete responders is quite recent and started to emerge just over the last 15 years. Although very few large retrospective studies or systematic reviews/meta-analyses have been published so far, results are still at an early stage, mostly because there are no robust markers predictive of pCR (molecular, clinical or radiological), a number of surgical approaches have been considered (from local excisions to abdominoperianel resection) and there is no consensus regarding the adjuvant treatment following surgical resection. However, the management of response following neoCHT-RT is the challenge of our times. A key issue in relation to pCR, is the presence of residual cancerous cells within lymph-nodes harvested in the surgical specimen (ypT0N+). These patients account for the 6.7-17.4% of ypT0 and are seldom analyzed. Nevertheless, literature published so far documented that a clinical nodal positivity before neoCHT-RT has been correlated with nodal metastases. An accurate prediction of the nodal status, however, would be crucial in order to tailor surgical choices. A number of pathways have been investigated including DNA repairs, apoptosis and growth signaling. Few studies investigated KRAS and p53 mutations, microRNAs', EGFR and VEGF expressions in relation to response, but despite the intensive research, results are quite scant. The most promising results came from studies using microarray technology, however, these studies have been conducted on a relative small number of patients and not always with a comparative purpose. Of note, a hallmark in the field of colorectal cancer (CRC) molecular profile is the consensus conducted that identified 4 cancer molecular subtypes (CMS) with distinct molecular features, classified as: MSI Immune, Canonical, Metabolic and Mesenchymal. It seems important to highlight that, since this classification has been just introduced, no one investigated ypT0N0/N+ patients in relation to the CMS sub-groups. Standard surgical approach for rectal cancer after neoCHT-RT include low anterior resection or abdominoperinal resection (if the sphincter is involved) with TME and an harvest of at least 12 nodes. Currently, a full thickness local excision (LE) can be proposed in high selected cases, if patients refuse a permanent stoma creation, if there are severe co-morbilities (patients unfit for major surgery) after a risk assessment of recurrences using validate criteria including nomograms. As expected, ypT0 patients have been reported with favorable outcomes, however, few issues need still to be delineated; however, survivals were not analyzed according to the ypT0-N status. Moreover, it has been reported that pCR did not show additional benefits from adjuvant chemotherapy with the endpoint of survivals, but ypT0N0/N+ were not stratified.

Preliminary Investigation. Dr Lorenzon is the PI of a preliminary study conducted on behalf of Italian Society of Surgical Oncology (SICO), young Board (YSICO) focused on ypT0 patients (Eur J Surg Oncol 2017;43:1472-1480). The study collected data of ypT0 patients treated at 13 centres (19 Italians and 2 Spanish) over the last 10 years independently from the neoCHT-RT performed, type of surgical approach or the nodal status. Each centre participated with a Y-SICO investigator (junior member) for data collection and a senior supervising member for mentorship and quality data validation. Dr Lorenzon analyzed data from 260 ypT0 patients (8.7% were ypT0N+). In line with the literature concerns, the majority of the patients did not perform adjuvant chemotherapy following surgery. At a mean follow-up of 47.6 months, 22 of the patients presented recurrences, 91% of them localized at distant site, mainly at the liver. Finally, results from uni/multivariate analyses documented that a nodal positivity was an independent variable correlated with survival. Although highly promising, these results should be further validated by a larger and powered analysis.

Study Rational and Hypothesis. So far, literature on ypT0 is encouraging but lacks of evidences. Accordingly, and on the basis of: A) The critical issues highlighted; B) The lack of validated features in particular regarding the ypT0N+ subgroup and C) The preliminary investigation and the impact that ypN+ had on survival, the rational of this study is to investigate a large number of ypT0 patients in relation to the nodal status, in order to define their clinical, radiological and molecular characteristics and to further validate survival outcomes. The two main hypotheses to test are whether we can distinguish ypT0N0 vs ypT0N+ and if the nodal positivity is a confirmed as an independent prognostic factor. Additionally, we will outline the pattern of recurrences and will assess the benefits and the compliance that these 2 groups have with adjuvant chemotherapy treatment. The results of this study would dramatically impact surgical and oncological choices for responders.

Specific Aim 1. To create a large Database of ypT0 patients from multiple institutions by involvement of young researchers (short-term aim) Specific Aim 2. To compare ypT0N0 vs ypT0N+ patients with respect of their clinical and molecular features (mid-term aim) Specific Aim 3. To define pattern and timing of relapses and to conduct a multivariate analysis of survivals which would include the N status and the use of adjuvant treatment (long-term aim) Methodology. The CORSiCA project is a multi-centre, multidisciplinary, observational study that will have a retrospective and a prospective line of research. The retrospective investigation will collect clinical, pathological and radiological data of patients >18 years with a final diagnosis of ypT0 in the surgical specimen treated over the last 5 years, independently from the neoCHT-RT performed (long course CHT-RT, short course RT), type of surgical resection (LE or TME) or nodal status. The prospective line of research will be conducted with the same inclusion criteria for 6 months plus 2 years of follow-up. Patients will be excluded if presenting with metastasis at diagnosis (clinical Stage IV), if treated exclusively with neo-adjuvant chemotherapy or if presenting peri-operative mortality.

Database creation (short term Aim 1). Clinical data will be acquired using a Database (DB). Patients' data will be uploaded anonymously in the DB with a consecutive number. Participants will be blinded to the other centres enrollment and exclusively the PI will be provided with the password for general data analysis. A case report form (eCRF) will be designed adhering to the quality standards in surgical research and in accordance with the STROBE Statement for collection, interpretation and divulgation of results. CRF will collect demographics (age, sex), tumoral features (distance from the anal verge, presence of stenosis, diameter), imaging staging modalities and assessment before and after neoCHT-RT (CT, MRI and PET scans), neoadjuvant scheme and radiation dose, weeks of interval to surgery, surgical procedures, peri-operative outcome (stoma creation, Clavien's co-morbility, hospital stay), pathologic data (mesorectal integrity, lymph node harvested, number of positive nodes, R status, pathologic N stage) and finally long term outcomes; also DICOM MRI and PET data will be uploaded for the further radiological analyses. Moreover, the availability of a pre-neoCHT-RT biopsy will be reported. Deliverables at this stage will include: DB design, study registration, centres recruitment and ethical board approval along with the starts of quality checks. Milestone: achievement of the 5 years of retrospective patients enrollment.

ypT0N0 vs ypT0N+ Sub-groups comparison (mid-term Aim 2). Patients presenting nodal positivity on TME specimens will be compared to the nodal negative patients for statistical purpose. Comparison will aim to define clinical, radiological and molecular features.

Statistics. ypT0N+ patients will be matched with ypT0N0 patients for statistical purpose using the propensity score matching method (PSM) and the following covariates: age, distance from the anal verge, clinical Stage, neoadjuvant approach. Continuous variables will be analyzed using means and standard deviations, whereas categorical variables will be analyzed using frequencies and percents. The groups will be compared using the T-test and Chi-square tests. All tests will be performed two-tailed and a p value <0.05 will be considered as statistically significant. A multivariate logistic regression will be performed with the end-point of nodal positivity (dependent variable) investigating the following putative independent variables: distance from the anal verge, tumor diameter, pre-treatment clinical stage (cT, cN, CRM), re-staging assessment (radiological major vs partial/absence of response), neo-adjuvant scheme (long-course CHT-RT vs short term RT). Although no limits of enrollment will be fixed for DB registration, we estimated power for 1000 patients uploaded, on the basis of the differences documented in the preliminary investigation, given an alpha error of 0.05. The computed calculation for a two-tailed T-test (independent groups) with an effect size of 0.3 estimated a power 1-beta of 0.811; on the other hand, both the computed calculations for a two-tailed Chi-square test with an effect size 0.01 and Kaplan Meier curves, estimated a power 1-beta>0.9. Statistical analyses will be obtained using SPSS Software and a bio-statistician will be enrolled for data analyses.

ypT0 vs ypT0N+ Molecular Analysis. Gene expression profiling (GEP) by microarray analysis will be performed using the NanoString nCounter Platform. Analyses will be conducted using the nCounter® PanCancer Progression Panel which can investigate 776 genes on a variety of sample types, including formalin-fixed paraffin-embedded (FFPE) tumor sections. Molecular GEP will be performed on FFPE tumoral endoscopic biopsies obtained before beginning of neo-adjuvant treatment of ypN+ patients matched by PSM with the ones obtained before neoCHT-RT of ypN0 patients; analyses will be conducted by a pathologist. FFPE biopsies will be transported from centres to the PI HI according to standard recommendations.

GEP power and Statistics. Given 776 genes of the Progression Panel, with 0.2 acceptable number of false positive, a desired fold difference of 1.8, a desired power of 0.9 and a standard deviation of 0.7, the investigation should be conducted on two groups of 35 patients. The correlation between genes expressions the clinical and pathological features of patients will be evaluated with the Spearman correlation coefficient also in relation to the CMS classification.

Deliverables of this stage will include: clinical, radiological and molecular analyses along with the quality data validation. Milestones: conclusion of the 6 months of prospective enrollment and the publication of mid-term results.

Oncological Outcome (long-term Aim 3). ypT0N0 patients and ypT0N+ patients will be compared with the end-points of overall survival (OS, any cause of death), disease free survival (DFS, first recurrence after surgical resection) and disease specific survival (DSS, death related to colorectal cancer) at 2 years of follow up, using the Kaplan Meier method; Cox regression model will investigate the impact that different variables (including nodal positivity and adjuvant treatment) have on survivals. We will evaluate also the quality of life of ypT0 patients using validated questionnaires. Data analyses will be conducted with a radiotherapist and an oncologist. Deliverables of this stage will include: survivals and quality of life analyses. Milestone: final analyses and publication of long-term results.

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer patients who underwent neo-adjuvant treatment followed by surgical resection
* Final pathologic diagnosis of absence of residual viable tumoral cells within the rectal wall specimen (pathologic complete response, pCR - ypT0).

Exclusion Criteria:

* Patients treated with chemotherapy-only protocols
* Stage IV
* Patients presenting peri-operative mortality (< 30 days from the surgical procedure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rectal cancer patients who underwent neo-adjuvant treatment followed by surgical resection with a final pathologic diagnosis of absence of residual viable tumoral cells within the rectal wall specimen (pathologic complete response, pCR - ypT0).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 24 months
  Any case of death

SECONDARY OUTCOMES:
Disease Free Survival | 24 months
  First recurrence after surgery
Disease Specific Survival | 24 months
  Death related to colorectal cancer
Molecular Profile of N+ | 24 months
  Molecular profiling of nodal positive patients (grant applied)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Lorenzon, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli
Locations (1):
- Fondazione Policlinico Unversitario Agostino Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) available to other researchers

REFERENCES:
- [Background] Ferlay J, Steliarova-Foucher E, Lortet-Tieulent J, Rosso S, Coebergh JW, Comber H, Forman D, Bray F. Cancer incidence and mortality patterns in Europe: estimates for 40 countries in 2012. Eur J Cancer. 2013 Apr;49(6):1374-403. doi: 10.1016/j.ejca.2012.12.027. Epub 2013 Feb 26. PMID 23485231
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] Heald RJ, Ryall RD. Recurrence and survival after total mesorectal excision for rectal cancer. Lancet. 1986 Jun 28;1(8496):1479-82. doi: 10.1016/s0140-6736(86)91510-2. PMID 2425199
- [Background] Kapiteijn E, Putter H, van de Velde CJ; Cooperative investigators of the Dutch ColoRectal Cancer Group. Impact of the introduction and training of total mesorectal excision on recurrence and survival in rectal cancer in The Netherlands. Br J Surg. 2002 Sep;89(9):1142-9. doi: 10.1046/j.1365-2168.2002.02196.x. PMID 12190680
- [Background] van Gijn W, Marijnen CA, Nagtegaal ID, Kranenbarg EM, Putter H, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer: 12-year follow-up of the multicentre, randomised controlled TME trial. Lancet Oncol. 2011 Jun;12(6):575-82. doi: 10.1016/S1470-2045(11)70097-3. Epub 2011 May 17. PMID 21596621
- [Background] Bujko K, Nowacki MP, Nasierowska-Guttmejer A, Michalski W, Bebenek M, Kryj M. Long-term results of a randomized trial comparing preoperative short-course radiotherapy with preoperative conventionally fractionated chemoradiation for rectal cancer. Br J Surg. 2006 Oct;93(10):1215-23. doi: 10.1002/bjs.5506. PMID 16983741
- [Background] Gerard JP, Conroy T, Bonnetain F, Bouche O, Chapet O, Closon-Dejardin MT, Untereiner M, Leduc B, Francois E, Maurel J, Seitz JF, Buecher B, Mackiewicz R, Ducreux M, Bedenne L. Preoperative radiotherapy with or without concurrent fluorouracil and leucovorin in T3-4 rectal cancers: results of FFCD 9203. J Clin Oncol. 2006 Oct 1;24(28):4620-5. doi: 10.1200/JCO.2006.06.7629. PMID 17008704
- [Background] Sauer R, Liersch T, Merkel S, Fietkau R, Hohenberger W, Hess C, Becker H, Raab HR, Villanueva MT, Witzigmann H, Wittekind C, Beissbarth T, Rodel C. Preoperative versus postoperative chemoradiotherapy for locally advanced rectal cancer: results of the German CAO/ARO/AIO-94 randomized phase III trial after a median follow-up of 11 years. J Clin Oncol. 2012 Jun 1;30(16):1926-33. doi: 10.1200/JCO.2011.40.1836. Epub 2012 Apr 23. PMID 22529255
- [Background] Bosset JF, Calais G, Mineur L, Maingon P, Stojanovic-Rundic S, Bensadoun RJ, Bardet E, Beny A, Ollier JC, Bolla M, Marchal D, Van Laethem JL, Klein V, Giralt J, Clavere P, Glanzmann C, Cellier P, Collette L; EORTC Radiation Oncology Group. Fluorouracil-based adjuvant chemotherapy after preoperative chemoradiotherapy in rectal cancer: long-term results of the EORTC 22921 randomised study. Lancet Oncol. 2014 Feb;15(2):184-90. doi: 10.1016/S1470-2045(13)70599-0. Epub 2014 Jan 17. PMID 24440473
- [Background] Schmoll HJ, Van Cutsem E, Stein A, Valentini V, Glimelius B, Haustermans K, Nordlinger B, van de Velde CJ, Balmana J, Regula J, Nagtegaal ID, Beets-Tan RG, Arnold D, Ciardiello F, Hoff P, Kerr D, Kohne CH, Labianca R, Price T, Scheithauer W, Sobrero A, Tabernero J, Aderka D, Barroso S, Bodoky G, Douillard JY, El Ghazaly H, Gallardo J, Garin A, Glynne-Jones R, Jordan K, Meshcheryakov A, Papamichail D, Pfeiffer P, Souglakos I, Turhal S, Cervantes A. ESMO Consensus Guidelines for management of patients with colon and rectal cancer. a personalized approach to clinical decision making. Ann Oncol. 2012 Oct;23(10):2479-2516. doi: 10.1093/annonc/mds236. PMID 23012255
- [Background] NCCN Clinical Practice Guidelines in Oncology (NCCN Guidelines®) Version 2.2016; 04.06.2016; www.nccn.org
- [Background] Habr-Gama A, Perez RO, Nadalin W, Sabbaga J, Ribeiro U Jr, Silva e Sousa AH Jr, Campos FG, Kiss DR, Gama-Rodrigues J. Operative versus nonoperative treatment for stage 0 distal rectal cancer following chemoradiation therapy: long-term results. Ann Surg. 2004 Oct;240(4):711-7; discussion 717-8. doi: 10.1097/01.sla.0000141194.27992.32. PMID 15383798
- [Background] Al-Sukhni E, Attwood K, Mattson DM, Gabriel E, Nurkin SJ. Predictors of Pathologic Complete Response Following Neoadjuvant Chemoradiotherapy for Rectal Cancer. Ann Surg Oncol. 2016 Apr;23(4):1177-86. doi: 10.1245/s10434-015-5017-y. Epub 2015 Dec 14. PMID 26668083
- [Background] Capirci C, Valentini V, Cionini L, De Paoli A, Rodel C, Glynne-Jones R, Coco C, Romano M, Mantello G, Palazzi S, Mattia FO, Friso ML, Genovesi D, Vidali C, Gambacorta MA, Buffoli A, Lupattelli M, Favretto MS, La Torre G. Prognostic value of pathologic complete response after neoadjuvant therapy in locally advanced rectal cancer: long-term analysis of 566 ypCR patients. Int J Radiat Oncol Biol Phys. 2008 Sep 1;72(1):99-107. doi: 10.1016/j.ijrobp.2007.12.019. Epub 2008 Apr 11. PMID 18407433
- [Background] Maas M, Nelemans PJ, Valentini V, Das P, Rodel C, Kuo LJ, Calvo FA, Garcia-Aguilar J, Glynne-Jones R, Haustermans K, Mohiuddin M, Pucciarelli S, Small W Jr, Suarez J, Theodoropoulos G, Biondo S, Beets-Tan RG, Beets GL. Long-term outcome in patients with a pathological complete response after chemoradiation for rectal cancer: a pooled analysis of individual patient data. Lancet Oncol. 2010 Sep;11(9):835-44. doi: 10.1016/S1470-2045(10)70172-8. Epub 2010 Aug 6. PMID 20692872
- [Background] Maas M, Nelemans PJ, Valentini V, Crane CH, Capirci C, Rodel C, Nash GM, Kuo LJ, Glynne-Jones R, Garcia-Aguilar J, Suarez J, Calvo FA, Pucciarelli S, Biondo S, Theodoropoulos G, Lambregts DM, Beets-Tan RG, Beets GL. Adjuvant chemotherapy in rectal cancer: defining subgroups who may benefit after neoadjuvant chemoradiation and resection: a pooled analysis of 3,313 patients. Int J Cancer. 2015 Jul 1;137(1):212-20. doi: 10.1002/ijc.29355. Epub 2014 Dec 13. PMID 25418551
- [Background] Probst CP, Becerra AZ, Aquina CT, Tejani MA, Wexner SD, Garcia-Aguilar J, Remzi FH, Dietz DW, Monson JR, Fleming FJ; Consortium for Optimizing the Surgical Treatment of Rectal Cancer (OSTRiCh). Extended Intervals after Neoadjuvant Therapy in Locally Advanced Rectal Cancer: The Key to Improved Tumor Response and Potential Organ Preservation. J Am Coll Surg. 2015 Aug;221(2):430-40. doi: 10.1016/j.jamcollsurg.2015.04.010. Epub 2015 Apr 23. PMID 26206642
- [Background] Martin ST, Heneghan HM, Winter DC. Systematic review and meta-analysis of outcomes following pathological complete response to neoadjuvant chemoradiotherapy for rectal cancer. Br J Surg. 2012 Jul;99(7):918-28. doi: 10.1002/bjs.8702. Epub 2012 Feb 23. PMID 22362002
- [Background] Ryan JE, Warrier SK, Lynch AC, Heriot AG. Assessing pathological complete response to neoadjuvant chemoradiotherapy in locally advanced rectal cancer: a systematic review. Colorectal Dis. 2015 Oct;17(10):849-61. doi: 10.1111/codi.13081. PMID 26260213
- [Background] Ryan JE, Warrier SK, Lynch AC, Ramsay RG, Phillips WA, Heriot AG. Predicting pathological complete response to neoadjuvant chemoradiotherapy in locally advanced rectal cancer: a systematic review. Colorectal Dis. 2016 Mar;18(3):234-46. doi: 10.1111/codi.13207. PMID 26531759
- [Background] Bosch SL, Vermeer TA, West NP, Swellengrebel HA, Marijnen CA, Cats A, Verhoef C, van Lijnschoten I, de Wilt JH, Rutten HJ, Nagtegaal ID. Clinicopathological characteristics predict lymph node metastases in ypT0-2 rectal cancer after chemoradiotherapy. Histopathology. 2016 Nov;69(5):839-848. doi: 10.1111/his.13008. Epub 2016 Jul 26. PMID 27270756
- [Background] Park IJ, You YN, Skibber JM, Rodriguez-Bigas MA, Feig B, Nguyen S, Hu CY, Chang GJ. Comparative analysis of lymph node metastases in patients with ypT0-2 rectal cancers after neoadjuvant chemoradiotherapy. Dis Colon Rectum. 2013 Feb;56(2):135-41. doi: 10.1097/DCR.0b013e318278ff8a. PMID 23303140
- [Background] Wan J, Liu K, Zhu J, Li G, Zhang Z. Implications for selecting local excision in locally advanced rectal cancer after preoperative chemoradiation. Oncotarget. 2015 May 10;6(13):11714-22. doi: 10.18632/oncotarget.3418. PMID 25909169
- [Background] Guinney J, Dienstmann R, Wang X, de Reynies A, Schlicker A, Soneson C, Marisa L, Roepman P, Nyamundanda G, Angelino P, Bot BM, Morris JS, Simon IM, Gerster S, Fessler E, De Sousa E Melo F, Missiaglia E, Ramay H, Barras D, Homicsko K, Maru D, Manyam GC, Broom B, Boige V, Perez-Villamil B, Laderas T, Salazar R, Gray JW, Hanahan D, Tabernero J, Bernards R, Friend SH, Laurent-Puig P, Medema JP, Sadanandam A, Wessels L, Delorenzi M, Kopetz S, Vermeulen L, Tejpar S. The consensus molecular subtypes of colorectal cancer. Nat Med. 2015 Nov;21(11):1350-6. doi: 10.1038/nm.3967. Epub 2015 Oct 12. PMID 26457759
- [Background] MERCURY Study Group. Diagnostic accuracy of preoperative magnetic resonance imaging in predicting curative resection of rectal cancer: prospective observational study. BMJ. 2006 Oct 14;333(7572):779. doi: 10.1136/bmj.38937.646400.55. Epub 2006 Sep 19. PMID 16984925
- [Background] Martens MH, van Heeswijk MM, van den Broek JJ, Rao SX, Vandecaveye V, Vliegen RA, Schreurs WH, Beets GL, Lambregts DM, Beets-Tan RG. Prospective, Multicenter Validation Study of Magnetic Resonance Volumetry for Response Assessment After Preoperative Chemoradiation in Rectal Cancer: Can the Results in the Literature be Reproduced? Int J Radiat Oncol Biol Phys. 2015 Dec 1;93(5):1005-14. doi: 10.1016/j.ijrobp.2015.09.008. Epub 2015 Sep 15. PMID 26581139
- [Background] McNair AG, Whistance RN, Forsythe RO, Macefield R, Rees J, Pullyblank AM, Avery KN, Brookes ST, Thomas MG, Sylvester PA, Russell A, Oliver A, Morton D, Kennedy R, Jayne DG, Huxtable R, Hackett R, Dutton SJ, Coleman MG, Card M, Brown J, Blazeby JM. Core Outcomes for Colorectal Cancer Surgery: A Consensus Study. PLoS Med. 2016 Aug 9;13(8):e1002071. doi: 10.1371/journal.pmed.1002071. eCollection 2016 Aug. PMID 27505051
- [Background] http://www.oncoguida.it/html//home.asp
- [Background] http://www.essoweb.org/eursso/quality-assurance/eurecca-project.html
- [Background] Tanis E, Caballero C, Collette L, Verleye L, den Dulk M, Lacombe D, Schuhmacher C, Werutsky G. The European Organization for Research and Treatment for Cancer (EORTC) strategy for quality assurance in surgical clinical research: Assessment of the past and moving towards the future. Eur J Surg Oncol. 2016 Aug;42(8):1115-22. doi: 10.1016/j.ejso.2016.04.052. Epub 2016 Apr 27. PMID 27241924
- [Background] Chia SK, Bramwell VH, Tu D, Shepherd LE, Jiang S, Vickery T, Mardis E, Leung S, Ung K, Pritchard KI, Parker JS, Bernard PS, Perou CM, Ellis MJ, Nielsen TO. A 50-gene intrinsic subtype classifier for prognosis and prediction of benefit from adjuvant tamoxifen. Clin Cancer Res. 2012 Aug 15;18(16):4465-72. doi: 10.1158/1078-0432.CCR-12-0286. Epub 2012 Jun 18. PMID 22711706
- [Background] http://strobe-statement.org
- [Background] Austin PC. A critical appraisal of propensity-score matching in the medical literature between 1996 and 2003. Stat Med. 2008 May 30;27(12):2037-49. doi: 10.1002/sim.3150. PMID 18038446
- [Background] Jandova J, Xu W, Nfonsam V. Sporadic early-onset colon cancer expresses unique molecular features. J Surg Res. 2016 Jul;204(1):251-60. doi: 10.1016/j.jss.2016.04.068. Epub 2016 May 6. PMID 27451894
- [Background] Chen X, Deane NG, Lewis KB, Li J, Zhu J, Washington MK, Beauchamp RD. Comparison of Nanostring nCounter(R) Data on FFPE Colon Cancer Samples and Affymetrix Microarray Data on Matched Frozen Tissues. PLoS One. 2016 May 13;11(5):e0153784. doi: 10.1371/journal.pone.0153784. eCollection 2016. PMID 27176004
- [Background] Veldman-Jones MH, Brant R, Rooney C, Geh C, Emery H, Harbron CG, Wappett M, Sharpe A, Dymond M, Barrett JC, Harrington EA, Marshall G. Evaluating Robustness and Sensitivity of the NanoString Technologies nCounter Platform to Enable Multiplexed Gene Expression Analysis of Clinical Samples. Cancer Res. 2015 Jul 1;75(13):2587-93. doi: 10.1158/0008-5472.CAN-15-0262. Epub 2015 Jun 11. PMID 26069246
- [Background] Ellervik C, Vaught J. Preanalytical variables affecting the integrity of human biospecimens in biobanking. Clin Chem. 2015 Jul;61(7):914-34. doi: 10.1373/clinchem.2014.228783. Epub 2015 May 15. PMID 25979952
- [Background] Department of Bioinformatics and Computational Biology, University of Texas MD Anderson Cancer Center, Houston, TX http://bioinformatics.mdanderson.org/MicroarraySampleSize/)
- [Background] Brown G, Richards CJ, Bourne MW, Newcombe RG, Radcliffe AG, Dallimore NS, Williams GT. Morphologic predictors of lymph node status in rectal cancer with use of high-spatial-resolution MR imaging with histopathologic comparison. Radiology. 2003 May;227(2):371-7. doi: 10.1148/radiol.2272011747. PMID 12732695
- [Background] Wilkins S, Haydon A, Porter I, Oliva K, Staples M, Carne P, McMurrick P, Bell S. Complete Pathological Response After Neoadjuvant Long-Course Chemoradiotherapy for Rectal Cancer and Its Relationship to the Degree of T3 Mesorectal Invasion. Dis Colon Rectum. 2016 May;59(5):361-8. doi: 10.1097/DCR.0000000000000564. PMID 27050597
- [Background] Gujral S, Conroy T, Fleissner C, Sezer O, King PM, Avery KN, Sylvester P, Koller M, Sprangers MA, Blazeby JM; European Organisation for Research and Treatment of Cancer Quality of Life Group. Assessing quality of life in patients with colorectal cancer: an update of the EORTC quality of life questionnaire. Eur J Cancer. 2007 Jul;43(10):1564-73. doi: 10.1016/j.ejca.2007.04.005. Epub 2007 May 22. PMID 17521904